CLINICAL TRIAL: NCT03351998
Title: Impact of Statin Therapy on Muscle Mitochondrial Function and Aerobic Capacity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Kansas Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00140789; R01AR071263 (NIH)
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-11

CONDITIONS: Mitochondrial Diseases
Keywords: insulin sensitivity; cardiorespiratory fitness; skeletal muscle mitochondrial function
MeSH Terms: conditions — Mitochondrial Diseases; Insulin Resistance | interventions — Atorvastatin; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Placebo (Placebo Comparator): Participants receiving matching placebo oral tablet.
  Interventions: Drug: Placebo Oral Tablet
- Low dose statin (Active Comparator): Participants will receive Lipitor 20Mg Tablet to take daily.
  Interventions: Drug: Lipitor 20Mg Tablet
- High dose statin (Active Comparator): Participants will receive Lipitor 80Mg Tablet to take daily.
  Interventions: Drug: Lipitor 80Mg Tablet

INTERVENTIONS:
Drug: Lipitor 20Mg Tablet — 20 mg/day pills.
  Other Names: atorvastatin
  Arms: Low dose statin
Drug: Lipitor 80Mg Tablet — 80 mg/day pills.
  Other Names: atorvastatin
  Arms: High dose statin
Drug: Placebo Oral Tablet — Matching placebo pill.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to test how different doses of a statin, Lipitor, affect muscle health and function, and cardiovascular fitness.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 25-43
* Weight stable (no more than 5% change in body weight the previous 3 months)
* >5% risk for a cardiovascular event in the next 10 years according to the 2013 American College of Cardiology/American Heart Association risk calculator and/or 2 out of 5 metabolic syndrome risk factors (Triglycerides ≥ 150 mg/dL; HDL ≤ 40 mg/dL; Glucose ≥ 100mg/dL; Waist Circumference ≥ 102cm for males, 88cm for females; Blood pressure: ≥ 130mmHg systolic and/or 85mmHg diastolic or being treated for hypertension) and/or LDL-Cholesterol >120 mg/dl.
* Stable doses of medications for 90 days
* Willing to stop all Nonsteroidal Antiinflammatory Drugs (NSAIDs) and aspirin for 7 days prior to muscle biopsy

Exclusion Criteria:

* Smoking
* Previous use of statins
* Use of other medications or supplements that affect lipid profiles or body weight in the last 6 months (e.g., fibric acids, bile acid sequestrants, nicotinic acids, fish oil)
* Diagnosis of chronic diseases including CVD, other metabolic diseases (e.g., thyroid), current diagnosis and active treatment of cancer, HIV, or acquired immunodeficiency syndrome.
* Diagnosis of type 1 or type 2 diabetes at the time of screening (fasting blood glucose >126mg/dL). If evidence of type 2 diabetes outcome measures is detected during the course of the study (fasting glucose > 126 mg/dl or HbA1c > 6.5%) we will notify the participant to contact their physician.
* History of abnormal bleeding problems
* Currently taking (within the last 10 days) anti-platelet medication (Plavix), Warfarin, and other anti-coagulants (eliquis, pradaxa, and xarelto) medications.
* >2 fold upper normal limit (UNL) for alanine aminotransferase (ALT) or creatinine
* Women who are pregnant or breastfeeding
* Individuals with polymorphisms (SLCO1B1 and GATM) known to be associated with susceptibility for statin induced myopathies (tested at screening)
* Currently enrolled in another research study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Thyfault, PhD, Principal Investigator — University of Kansas Medical Center
Locations (2):
- United States (2):
  - University of Kansas Medical Center, Kansas City, Kansas
  - East Carolina University, Greenville, North Carolina

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All 68 participants that were officially enrolled were randomized.
Period: Overall Study
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
Started | 23 | 24 | 21
Completed | 16 | 19 | 17
Not Completed | 7 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose Statin | High Dose Statin | Total
Number analyzed (Participants) | 23 | 24 | 21 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.98 (8.28) | 54.53 (7.66) | 54.10 (7.14) | 53.87 (7.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 16 | 49
  Male | 7 | 7 | 5 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 3 | 6
  White | 20 | 23 | 16 | 59
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 23 | 24 | 21 | 68
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 199.65 (38.82) | 211.75 (41.68) | 214.33 (33.53) | 208 (38.32)
Weight [Mean (Standard Deviation); unit: kg] | 93.79 (13.89) | 90.60 (15.87) | 89.28 (15.22) | 91.27 (14.92)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 32.96 (4.55) | 31.14 (3.74) | 32.31 (4.98) | 32.12 (4.43)
Relative Peak VO2 Max [Mean (Standard Deviation); unit: mL/kg/min] | 24.12 (5.7) | 25.53 (6.97) | 24.92 (5.12) | 24.87 (5.96)

OUTCOME MEASURES:

1. Primary Outcome: Difference in Mitochondrial Respiratory Function
Time Frame: value at 12 months minus value at baseline
Measure: Mean (Standard Deviation); unit: pmols/s/mg
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
Number analyzed (Participants) | 16 | 17 | 16
pmols/s/mg | 36 (366) | 32 (213) | -3 (180)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.6051, signed rank test; This is within group 12 month change; Mean Difference (Net) = 36.02, Standard Deviation 365.55
Statistical Analysis 2: Comparison: Low Dose Statin; Test type: Superiority; p = 0.9434, signed rank test; This is within group 12 month change; Mean Difference (Net) = 31.89, Standard Deviation 213
Statistical Analysis 3: Comparison: High Dose Statin; Test type: Superiority; p = 0.9408, t-test, 2 sided; This is within group 12 month change; Mean Difference (Net) = -3.39, Standard Deviation 179.54

2. Secondary Outcome: Change in VO2 Max
Time Frame: value at 12 months minus value at baseline
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
Number analyzed (Participants) | 15 | 18 | 17
L/min | -0.2 (0.23) | 0.03 (0.16) | -0.06 (0.18)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.7458, t-test, 2 sided; This is within group 12 month change; Mean Difference (Net) = -0.2, Standard Deviation 0.23
Statistical Analysis 2: Comparison: Low Dose Statin; Test type: Superiority; p = 0.4056, t-test, 2 sided; This is within group 12 month change; Mean Difference (Net) = 0.03, Standard Deviation 0.16
Statistical Analysis 3: Comparison: High Dose Statin; Test type: Superiority; p = 0.1932, t-test, 2 sided; This is within group 12 month change; Mean Difference (Net) = -0.06, Standard Deviation 0.18

ADVERSE EVENTS:
Time Frame: Participants were contacted weekly by phone or email and prompted to disclose any adverse events. Additional adverse events could be reported if participant contacted study team outside of the usual weekly check in. Adverse events were monitored until symptoms subsided or adverse event ended or until the end of the 12 month intervention period.
Description: The definitions used for adverse events and/or serious adverse events are the same as clinicaltrials.gov definitions
Arm/Group | Placebo | Low Dose Statin | High Dose Statin
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 1/23 | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 15/23 | 17/24 | 14/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Low Dose Statin (N=24) | High Dose Statin (N=21)
Cardiovascular event (SVT) unrelated to intervention (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Participant was diagnosed with an SVT that required hospitalization.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=23) | Low Dose Statin (N=24) | High Dose Statin (N=21)
COVID-19 (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 3 (3) | 0 (0)
UTI (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
GI Upset (Gastrointestinal disorders) | 2 (2) | 3 (3) | 3 (3)
Muscle or Joint Pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 8 (9) | 6 (7)
Adverse event related to testing for study (Investigations) | 2 (2) | 5 (6) | 2 (2) — Any mild to moderate adverse reaction to the testing procedures for the study. Examples include vein irritation after IVGTT, bruise or swelling at biopsy site.
Sinus Infection/Flu Symptoms (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3) | 3 (3)

LIMITATIONS AND CAVEATS:
The COVID-19 epidemic started in the middle of the trial forcing us to stop recruitment for four months. Furthermore, the continuation of the pandemic slowed recruitment for the rest of the trial and significantly impacted n size. There was also a national dextrose shortage following a hurricane in Puerto Rico. As a result many of the IVGTT were not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT03351998/Prot_SAP_000.pdf